CLINICAL TRIAL: NCT06342011
Title: Effects of Anti-inflammatory Diet on Inflammatory Markers, Anxiety, Depression and Quality of Life in Patients With Inflammatory Bowel Disease
Brief Title: Effect of Anti-inflammatory Diet in Patients With Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KY-2024-039
Record Dates: First submitted 2024-03-10; First posted 2024-04-02 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Anti-inflammatory diet; Inflammatory index; Quality of life
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular diet group (No Intervention): Explain disease related knowledge; According to the patient's situation, give personalized dietary guidance, establish regular eating habits, carefully evaluate the types of food in the food, and avoid spicy stimulation, gas production, high fat and other foods that are easy to cause intestinal discomfort. SMS follow-up was conducted 3 days after discharge, and weekly phone follow-up was conducted to see if patients needed to solve problems and help them solve them in time.
- Anti-inflammatory diet group (Experimental): AID knowledge education was given to patients in the intervention group after admission. At the same time, patients are asked to pay attention to the "anti-inflammatory diet" wechat mini program developed by researchers, and teach patients how to use it, including the choice of anti-inflammatory diet, inappropriate anti-inflammatory diet, diet alarm clock, diet notes and other related functions. Missionary patients persisted with AID until re-examination 8 weeks later.
  The researchers conducted weekly telephone follow-up to urge the patients to adhere to the AID diet, answer the questions raised by the patients during the implementation process, and understand the patients' knowledge acceptance and diet implementation. Follow-up is carried out by qualified members of the training research team. Follow-up can take the form of face-to-face visit to the community or direct telephone follow-up, and make follow-up records.
  Interventions: Behavioral: Anti-inflammatory diet group

INTERVENTIONS:
Behavioral: Anti-inflammatory diet group — Patients in the intervention group were given AID knowledge education, and patients were asked to pay attention to the "anti-inflammatory diet" wechat mini program developed by the researchers to teach patients how to use it, including the selection of anti-inflammatory diet, unsuitable anti-inflammatory diet, diet alarm clock, diet notes and other related functions. The missionary patients insisted on AID until reexamination 8 weeks later.
  Arms: Anti-inflammatory diet group

SUMMARY:
For the first time, this study developed an anti-inflammatory diet （AID） recipe suitable for Inflammatory bowel disease（IBD） patients and developed an AID application program to verify the intervention effect of AID on IBD patients, which not only promoted the application of AID in IBD patients and promoted the promotion of AID model, but also provided new ideas for the prevention and treatment strategies for IBD patients.

DETAILED DESCRIPTION:
This study aims to verify the intervention effect of AID on IBD patients, promote the promotion of AID model, and provide new ideas for the prevention and treatment strategies of IBD patients.

In this study, 66 IBD patients who met the inclusion criteria were divided into experimental group and control group by randomized controlled trial method. The experimental group was based on routine nursing measures, and the intervention group taught patients to take anti-inflammatory diet and use the anti-inflammatory diet mini-program developed by the researcher, daily anti-inflammatory diet, intervention time was 8 weeks, and observed the inflammatory indicators (white blood cells, neutrophils, erythrocyte precipitation, CRP), quality of life, anxiety and depression, self-efficacy and other conditions in the blood results of the patients before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of inflammatory bowel disease, the diagnostic criteria refer to the 2018 revised Consensus opinion on the diagnosis and treatment of inflammatory bowel disease;
2. The patient has clear consciousness and certain understanding, language expression and writing ability;
3. Patients participated in this study knowingly and voluntarily;
4. At least 18 years old.

Exclusion Criteria:

1. cognitive impairment, mental illness, accompanied by mental disorders;
2. Alcohol and drug abusers.
3. The patient could not participate in the researcher due to the deterioration of the condition;
4. Patients who voluntarily quit due to other reasons;
5. Those who did not complete the assessment scale during the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein | 8 weeks after intervention
  C-reactive protein (mg/L) is a non-specific inflammatory marker. It is an acute phase reaction protein synthesized by the liver to protect the body when pathogenic microorganisms invade the body.
Erythrocyte sedimentation rate (ESR) | 8 weeks after intervention
  Erythrocyte sedimentation rate (mm/h) refers to the rate of erythrocyte sedimentation under certain conditions. The anticoagulant blood is placed in a vertically erected small glass tube. Due to the large proportion of red blood cells, it is naturally sunk by gravity. Under normal circumstances, the subsidence is very slow. The rate of erythrocyte sedimentation is often expressed by the distance of red blood cells sinking at the end of the first hour, called ESR.
Leukocyte | 8 weeks after intervention
  White blood cells are colorless, spherical, nucleated blood cells. The total number of normal adults is (4.0 ~ 10.0)x 109/L, which can change in a certain range depending on the time of day and the functional state of the body.

SECONDARY OUTCOMES:
Self-Rating Anxiety Scale，SAS | 8 weeks after intervention
  This table, compiled by Zung in 1971, is used in SAS for a total of 20 symptom categories, with a score of 1 to 4 after each problem. The scoring scale is: "1" indicates that the symptom is rarely present; A score of "2" indicates that this symptom is sometimes present; A score of "3" indicates that the symptoms are present most of the time; A score of "4" indicates symptoms most of the time. The cut-off value of SAS standard score is 50 points, of which < 50 is no anxiety, 50 to 59 is mild anxiety, 60 to 69 is moderate anxiety, and more than 70 is severe anxiety.
Self-Rating depression scale，SDS | 8 weeks after intervention
  The scale is scored on the following scale: "1" means that this symptom rarely occurs; A score of "2" indicates that this symptom sometimes occurs; A score of "3" means the symptoms are present most of the time; A score of "4" means that symptoms occur in most cases. Among them, 10 items are positive (1, 2, 3, 4 points in sequence), and 2, 5, 6, 11, 12, 14, 16, 17, 18, 20 items are negative (4, 3, 2, 1 points in sequence). The total score is obtained by adding all the scores together. Multiply the total score by 1.25, and the points portion is obtained from the SDS standard score. SDS standard score 53 points, mild depression 53 to 62 points, moderate depression 63 to 72 points. Major depressive disorder is... Seventy-two o 'clock.
Simplified Chinese version of Inflammatory Bowel Disease Quality of Life Scale (IBDQ) | 8 weeks after intervention
  In this study, the simplified Chinese version of inflammatory bowel Disease Quality of Life Scale was used to assess the quality of life of IBD patients. This scale is the most widely used inflammatory bowel disease specific quality of life scale in the world, with a Cronbach's of 0.986, indicating good reliability and validity. The scale consists of 32 items and 4 dimensions, and mainly evaluates the intestinal symptoms, systemic symptoms, emotional ability and social ability of IBD patients. Each entry has seven options on a scale of 1-7, with 1 representing the worst and 7 representing the best, on a scale of 32-224, with higher scores indicating better quality of life.
Inflammatory Bowel Disease Self-Efficacy Scale (IBD-SES) | 8 weeks after intervention
  In this study, the Chinese version of the inflammatory bowel disease Self-efficacy Scale (GSES) was used for assessment. The GSES has 29 items and 4 dimensions, including stress and emotion management, medical care management, disease management and remission maintenance management. Cronbach's coefficient ranges from 0.899 to 0.973, and Guttman's half coefficient ranges from 0.825 to 0.917. Score using the Likert 10-level scoring method, with a total score of 29-290, the higher the score, the stronger the sense of self-efficacy.
Body Mass Index | 8 weeks after intervention
  The patient's weight gain was measured first，weight in kilograms, height in meters,weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Qian, BA, Principal Investigator — The Fourth Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No